CLINICAL TRIAL: NCT06706310
Title: Evaluate TQ-A3334 Tablets Combined Nucleoside (Acid) Analogs in the Initial Treatment/Chronic Hepatitis B Virus (HBV) Infection Subjects of Chronic HBV Infection
Brief Title: Evaluate TQ-A3334 Combined Nucleoside (Acid) Analogs in the First Treatment/Treatment of Chronic HBV Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ-A3334-II-03
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleosides; Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TQ-A3334 tablets 0.2mg quaque die (QD), combined with nucleoside (acid) analogs (NAs) (Active Comparator): TQA3334 tablets 0.2mg once a day 0.2 mg/time, 1 time/night, 48 weeks of administration; 1 time/day for combined medication, 72 weeks of administration; 72 weeks.
  Interventions: Drug: TQA3334 Tablet; Drug: Nucleoside (acid) analogs (NAs)
- 0.2mg quaque die (QD) placebo, combined with nucleoside (acid) analogs (NAs) (Placebo Comparator): Placebo tablets 0.2mg once a day,0.2 mg/time, 1 time/night, 48 weeks of administration; 1 time/day for combined medication, 72 weeks of administration; 72 weeks.
  Interventions: Drug: Placebo; Drug: Nucleoside (acid) analogs (NAs)
- TQ-A3334 tablets 0.5mg once the next day(QOD), combined with nucleoside (acid) analogs (NAs) (Active Comparator): TQA333 tablets 0.5mg once the next day once the next day, administration for 48 weeks; combined medication 1/day, 72 weeks of administration.
  Interventions: Drug: TQA3334 Tablet; Drug: Nucleoside (acid) analogs (NAs)
- Placebo 0.5mg once the next day (QOD) , combined with nucleoside (acid) analogs (NAs) (Placebo Comparator): Placebo 0.5mg once the next day, administration for 48 weeks; combined medication 1/day, 72 weeks of administration;
  Interventions: Drug: Placebo; Drug: Nucleoside (acid) analogs (NAs)
- TQ-A3334 tablets 0.5mg quaque die (QD), combined with nucleoside (acid) analogs (NAs) (Active Comparator): TQA3334 tablets 0.5mg once a day, 1/night, 48 weeks of administration; 1 time/day for combined medication, 72 weeks of administration; 72 weeks.
  Interventions: Drug: TQA3334 Tablet; Drug: Nucleoside (acid) analogs (NAs)
- Placebo 0.5mg quaque die (QD) combined with nucleoside (acid) analogs (NAs) (Placebo Comparator): Placebo 0.5mg once a day, 1/night, 48 weeks of administration; 1 time/day for combined medication, 72 weeks of administration; 72 weeks.
  Interventions: Drug: Placebo; Drug: Nucleoside (acid) analogs (NAs)

INTERVENTIONS:
Drug: Placebo — Placebo contains no active substance.
  Arms: 0.2mg quaque die (QD) placebo, combined with nucleoside (acid) analogs (NAs); Placebo 0.5mg once the next day (QOD) , combined with nucleoside (acid) analogs (NAs); Placebo 0.5mg quaque die (QD) combined with nucleoside (acid) analogs (NAs)
Drug: TQA3334 Tablet — Inhibit viral replication.
  Arms: TQ-A3334 tablets 0.2mg quaque die (QD), combined with nucleoside (acid) analogs (NAs); TQ-A3334 tablets 0.5mg once the next day(QOD), combined with nucleoside (acid) analogs (NAs); TQ-A3334 tablets 0.5mg quaque die (QD), combined with nucleoside (acid) analogs (NAs)
Drug: Nucleoside (acid) analogs (NAs) — Inhibit viral replication.

SUMMARY:
This study uses random, double -blindness, placebo control, and phase multi -center test design. All subjects who meet the standards receive TQ-A3334 per tablet/placebo nucleoside (acid) analog. A total of 116 subjects are needed.

ELIGIBILITY:
Inclusion Criteria:

Those who meet all the selected standards below can enter the group test:

* The subject can communicate well with the researchers and understand and comply with the various items in this study, understand and sign the consent of informed consent;
* 18-65 years old (including the boundary value), and men and women are not limited (calculated based on the date of signing the consent of informedness);
* Serum virus standard: serum HBSAG positive for more than 6 months or more than 6 months chronic Evidence of HBV infection.
* No obvious liver cirrhosis is judged by researchers;

Those who have been treated after treatment need to meet the following conditions:

* The subject must receive oral nucleoside (acid) drug treatment before screening ≥6 months and the stable treatment plan before the screening period is ≥3 months;
* Historian history records of the HBV DNA <6 and above HBV DNA <6) HBV DNA <minimum detection lower limit.

The initial governance subjects need to meet the following conditions:

* If the preliminary governance subject does not have HBSAG positive for 6 months, researchers can make the knot according to the initial diagnosis Fruit, the clinical manifestations of the subjects, and the comprehensive judgment of the family history of hepatitis B family whether it is chronic infection;
* The subjects have never received the treatment of chronic hepatitis B antiviral treatment (oral nucleoside drugs and interferon) at the time of screening;
* The upper limit of the normal reference value (ULN) <Alanine aminotransferase≤ 5 × ULN (within 2 weeks before the first medication)

Exclusion Criteria:

Anyone who appears below will not be able to enter the group test:

* Pregnancy (pregnancy test is positive) or lactating women.
* Combined other virus infections such as hepatitis A virus，hepatitis C virus, hepatitis D virus, hepatitis E virus, human immunodeficiency virus, syphilis (those with positive syphilis antibodies, and those who are judged by researchers) and so on.
* History of liver cirrhosis or before screening/screening shows significant fibrosis or liver cirrhosis; or abdominal ultrasound examination prompts suspected liver cirrhosis; past liver dysfunction history or screening period has liver dysfunction compensation For those such as ascites, hepatic brain diseases, and esophageal stomach veins, bleeding;
* The subject of Hepatocellular Carcinoma (HCC) before screening or at the time of screening has a history of Hepatocellular Carcinoma (HCC), or suspected HCC;
* There is a history of malignant tumor diseases within the first 5 years of screening. Except for specific menstrual resection, it can be completely cured (such as skin basal cell carcinoma, etc.).
* A subject with other chronic liver diseases, including but not limited to autoimmune liver disease, alcoholic liver disease, hepatolenticular degeneration, etc.
* Organization and bone marrow transplantation have been accepted in the past.
* Poor thyroid disease, or clinical thyroid dysfunction (TSH abnormal T3 or T4 abnormalities);
* Eye disease: Including the bottom of the eye lesions (changes in the cotton samples with symptoms of the eye) and retinal lesions.
* Autoimmune diseases include but are not limited to: systemic lupus erythematosus, rheumatoid arthritis, etc.
* In addition to liver disease, there are obvious systemic or major diseases.
* Any systemic anti -tumor (including radiation) or immunosuppressive treatment (including biomorphic inhibitors), or immunotherapies within 6 months before screening.
* Blood transfusion within ≤ 2 months before screening and/or donate blood within 1 month before screening. Note: The subject must not donate blood during the entire study;
* History of allergies to test medicines or its auxiliary materials;
* Toll-like receptors-7, Toll-like receptors-8 receptor agonist or PD-1, PD-L1 similar drugs have been used within three months before screening.
* The subject has participated in a clinical trial and accepted the test medicine for the test before the first time of the administration: 5 semi -half -life (such as known) or studying the duration of the biological effects (such as such as the duration of the biological effects (such as such as the duration of the biological effects (such as such as the duration of the biological effects (such as such as the duration of the biological effects (such as such as the duration of the biological effects (such as such as the duration of the biological effects (such as the duration of the biological effects (such as the duration of the biological effects (such as the duration of the biological effects (such as Two times (known) or 90 days (if the elderly prevails) or 90 days (if the half -life or duration is unknown).
* History or condition of cardiovascular disease: History of risk factors for risk factors of cutting -out rooms, including miracles, known long QT syndrome, heart failure, myocardial infarction, angina pectoris, or clinical significance laboratory Examination (including hypokalemia, hypercalcemia, or hypomagnesemia). Long QT syndrome or BRUGADA syndrome family history. ECG shows abnormal clinical significance. Heart rate≤45 Secondary/minutes.
* Researchers believe that those should not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
At 24 weeks, the changes in serum HBSAG relative to the baseline | Up to 24 weeks
  Evaluate the subject of chronic HBV infection in the early treatment/treatment of chronic HBV infection, TQ-A3334 combined with oral nucleoside (acid) drugs comparative placebo and oral nucleoside (acid) drugs, can it significantly improve the treatment for 24 weeks Serum HBSAG relative to the changes in the baseline

SECONDARY OUTCOMES:
The incidence of adverse events（AEs） | Up to 48 weeks
  To investigate the incidence of adverse events (AEs) during treatment
Severity of adverse events (AEs) | Up to 48 weeks
  To study the severity of adverse events (AEs) during treatment
Incidence of serious adverse events (SAEs) | Up to 48 weeks
  To investigate the incidence of serious adverse events (SAEs) during treatment
Severity of serious adverse events（SAEs） | Up to 28 weeks
  To investigate the severity of serious adverse events (SAEs) during treatment
HBsAg<100 IU/ml and HBV DNA <20 IU/ml subject | Week 24, 48 weeks, 60 weeks, 72 weeks
  The proportion of subjects of HBsAg<100 IU/ml and HBV DNA <20 IU/ml.
HBSAG self -based lines drop ≥0.5, ≥1 Log10IU/ml | Week 24, 48 weeks, 60 weeks, 72 weeks
  Awarded by HBSAG's self -base line decrease ≥0.5, ≥1 Log10IU/ml.
The proportion of subjects of HBSAG serological removal and/or serum transformation during the study period | Week 24, 48 weeks, 60 weeks, 72 weeks
  HBSAG serum science clearance and/or serum transition ratio proportion
The proportion of subjects of HBEAG serological removal and/or serum conversion during the study period | Week 24, 48 weeks, 60 weeks, 72 weeks
  The proportion of subjects of HBEAG serological removal and/or serum transformation during the study.
Peak time (Tmax) | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  Time to peak blood concentration after a single dose.
Peak Concentration | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  The highest plasma drug concentration that can be achieved after medication.
Area under blood concentration-time curve (AUC) | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  The amount of drug absorbed into the human circulation after a single dose can be estimated using the area under the blood concentration-time curve.
Apparent volume of distribution (Vd/F) | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  When a drug reaches homeostasis in the body, the ratio of the amount of drug in the body to the blood concentration is called the apparent volume of distribution
Plasma clearance | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, D15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, D57 and D85 0hour pre-dose.
  How many milliliters of plasma can the kidneys completely clear in unit time (per minute)
Elimination half-life time | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  The time it takes for the plasma concentration to drop by half.
Peaking Time | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, D15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, D57 and D85 0hour pre-dose.
  The time required to reach peak steady-state concentration after administration.
Steady state maximum concentration | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  The highest blood concentration that occurs after stabilization.
Steady state minimal concentration | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  The lowest blood concentration that occurs after stabilization
Area under steady-state blood concentration-time curve | Day1 0 hour pre-dose,10,20,30minutes,1,2,3,6,12,24,48 hours after dose, Day15 within 60 minutes pre-dose, Day29 0h pre-dose,10, 20, 30 minutes, 1,2,3,6,12,24,48 hours after dose, Day57 and Day85 0hour pre-dose
  After the dosage of a single agent, the amount of dosage of the blood circulation of the person can be used with blood concentration-the area of the area under the time curve.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Hospital workers in Liuzhou, Liuchow, Guangxi
  - WuHan Jinyintan Hospital, Wuhan, Hubei
  - The Second XIANGYA Hospital Of Central South University, Changsha, Hunan
  - The Fifth People's Hospital of Wuxi (Affiliated Wuxi Fifth Hospital of Jiangnan University), Wuxi, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Pu'er People's Hospital, Pu'er, Yunnan
  - People's Hospital Of RuiAn City, Rui’an, Zhejiang